CLINICAL TRIAL: NCT06655766
Title: Socket Preservation Using Socket-plug Technique With Alloplastic Putty Bone Versus Ice Cream Cone Technique in Extraction Socket With Buccal Dehiscence: A Randomized Controlled Clinical Trial.
Brief Title: Socket Preservation Using Socket-plug Technique With Alloplastic Putty Bone Versus Ice Cream Cone Technique in Extraction Socket With Buccal Dehiscence.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelrahman Medhat, Teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PER6-3-1 ..
Record Dates: First submitted 2024-10-20; First posted 2024-10-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Socket Preservation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Socket-plug technique with putty bone (Experimental): * Patients will be anesthetized at the surgical site by infiltration, using Articaine Hydrochloride 4%.
  * Atraumatic extractions after careful surgical preparation of the soft and hard tissues using periotomes sulcular incision may be done with the aid of number 15c scalpel to dissect the crestal fibers and avoid trauma to soft tissue, care should be taken not to raise the flap.
  * Careful curettage and debridement of the socket is performed with hand instruments to remove granulation tissue.
  * The socket walls are then inspected for the presence of buccal defects.
  * putty bone is injected into the socket up to the crest of the bone.
  * Collagen plug or sponge is adapted over the graft to occlude the socket
  * The plug is then stabilized with absorbable suture material.
  Interventions: Procedure: socket-plug technique with putty bone
- Ice cream cone technique (Active Comparator): * Patients will be anesthetized at the surgical site by infiltration, using Articaine Hydrochloride 4%.
  * Atraumatic extractions after careful surgical preparation of the soft and hard tissues using periotomes sulcular incision may be done with the aid of number 15c scalpel to dissect the crestal fibers and avoid trauma to soft tissue, care should be taken not to raise the flap.
  * Careful curettage and debridement of the socket is performed with hand instruments to remove granulation tissue.
  * The socket walls are then inspected for the presence of buccal defects.
  * A Collagen barrier membrane is then shaped as an ice-cream cone and placed in the extraction socket lining the buccal tissues.
  * The socket is then filled with particulate bone graft.
  * The upper part of the membrane is then used to cover the socket.
  * Absorbable suture is then used to close the socket and stabilize the barrier membrane
  Interventions: Procedure: Ice cream cone technique

INTERVENTIONS:
Procedure: socket-plug technique with putty bone — * Atraumatic extractions after careful surgical preparation of the soft and hard tissues using periotomes sulcular incision may be done with the aid of number 15c scalpel to dissect the crestal fibers and avoid trauma to soft tissue, care should be taken not to raise the flap.
  * Careful curettage and debridement of the socket is performed with hand instruments to remove granulation tissue.
  * The socket walls are then inspected for the presence of buccal defects.
  * putty bone is injected into the socket up to the crest of the bone.
  * Collagen plug or sponge is adapted over the graft to occlude the socket
  * The plug is then stabilized with absorbable suture material.
  Arms: Socket-plug technique with putty bone
Procedure: Ice cream cone technique — * Atraumatic extractions after careful surgical preparation of the soft and hard tissues using periotomes sulcular incision may be done with the aid of number 15c scalpel to dissect the crestal fibers and avoid trauma to soft tissue, care should be taken not to raise the flap.
  * Careful curettage and debridement of the socket is performed with hand instruments to remove granulation tissue.
  * The socket walls are then inspected for the presence of buccal defects.
  * A Collagen barrier membrane is then shaped as an ice-cream cone and placed in the extraction socket lining the buccal tissues.
  * The socket is then filled with particulate bone graft.
  * The upper part of the membrane is then used to cover the socket.
  * Absorbable suture is then used to close the socket and stabilize the barrier membrane
  Arms: Ice cream cone technique

SUMMARY:
Socket Preservation Using Socket-plug Technique with Alloplastic Putty Bone Versus Ice Cream Cone Technique in Extraction Socket with Buccal Dehiscence: A Randomized Controlled Clinical Trial.

DETAILED DESCRIPTION:
this randomized controlled clinical trial evaluates the effect of using alloplastic putty bone with socket-plug technique versus ice-cream cone technique regarding dimensional changes in bone width

ELIGIBILITY:
Inclusion Criteria:

* Single or double rooted teeth indicated for extraction.
* Systemically free patient
* Presence of small buccal dehiscence not exceeding 1/3 of the root.
* Maxillary and Mandibular Arches
* Non-smoker
* Adults or above the age of 21.
* Able to tolerate surgical periodontal procedures.
* Full mouth plaque and bleeding scores less than 15%.
* Compliance with the maintenance program.
* Provide informed consent

Exclusion Criteria:

* Systemic conditions/disease that contraindicate surgical procedure.
* Patients with presence or history of osteonecrosis of the jaws, with use of bisphosphonates, exposure to head and neck radiation, chemotherapy.
* Extraction socket with intact walls with no buccal dehiscence
* Patients with large distinct pre-apical pathology
* Heavy Smokers more than 10 cigarettes a day
* Patients without availability to attend follow-up visits or patients rejecting to sign the informed consent.
* Patients with parafunctional habits that produce overload on implant, such as bruxism and clenching.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2025-11-13 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative volumetric changes | day 0 - month 6
  Bone volumetric changes will be measured in millimeter by super-imposition of 3D scans using volume analysis software.

SECONDARY OUTCOMES:
Horizontal alveolar ridge width | day 0 - month 6
  Buccolingual alveolar ridge width will be measured in millimeter 1, 3, 5 mm bellow alveolar crest in both groups.
Vertical alveolar ridge height | day 0 - month 6
  Vertical alveolar ridge height will be measured in millimeter from the end of the socket to the alveolar crest in both groups.